CLINICAL TRIAL: NCT06066801
Title: Bedside Bone Biopsy Versus Conventional Bone Biopsy for Management of Diabetic Foot Osteomyelitis: an Open-label Controlled Randomized Non-inferiority Trial
Brief Title: Bedside Bone Biopsy in Diabetic Foot Osteomyelitis
Acronym: BOLBOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PHRC-21-0179; 2022-A02754-39 (Other: IDRCB)
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Subjects With Diabetes and DFU With a Suspicion of DFO
Keywords: Bedside bone biopsy, conventional bone biopsy, diabetes, Diabetic Foot Ulcer (DFU), diabetic foot osteomyelitis (DFO)
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bedside blind bone biopsy procedure (Experimental): Bedside blind bone biopsy procedure performed by a physician of the participating center through healthy skin with bone trocar following local and light systemic anesthesia. Samples will be analyzed for microbiology and histopathology
  Interventions: Procedure: Bedside blind bone biopsy procedure
- Standard bone biopsy procedure (Active Comparator): Standard BB procedure (surgical or radiological) performed according to the local standard of care of each participating center and done through healthy skin and under locoregional anesthesia. Samples will be analyzed for microbiology and histopathology
  Interventions: Procedure: Bedside blind bone biopsy procedure

INTERVENTIONS:
Procedure: Bedside blind bone biopsy procedure — It was performed in the patient's room under aseptic conditions. Pain relievers were given orally within the hour preceding the procedure. Superficial anesthesia was performed firstly subcutaneously and then on the periosteum, Inhaled anesthesia was started concomitantly. Following a short incision with a scalpel, the trocar inside a cannula was inserted through healthy skin at a minimum distance of 2 cm from the ulcer edge, close to the bone, preferentially on dorsal foot side. When the trocar was firmly inserted into the bone, it was pulled out from the cannula. Biopsy needle was then slipped into the cannula and twisted into the bone clockwise. Biopsy needle was then pulled out and the bone was pushed out with the ejector pin into a sterile surgical drape and divided in two parts.

SUMMARY:
During their lifetime, 15 to 25% of patients with diabetes mellitus will develop a Diabetic Foot Ulcer (DFU) related to neuropathy and/or peripheral arterial disease. DFU is the leading cause of non-traumatic lower-extremity amputation worldwide. Diabetic foot osteomyelitis (DFO), which complicates up to 60% of DFU, is a major trigger of amputation in over 80% of persons with diabetes resulting in subsequent loss of quality of life. It has been shown that medical treatment of DFO may prevent amputations with early diagnosis of osteomyelitis and appropriate use of antibiotics. Empirical antimicrobial treatment is not recommended for DFO as for other chronic infections. Surgically or radiologically acquired bone sample for culture is the reference standard recommended by the International Working Group of Diabetic Foot (IWGDF) to diagnose DFO and to determine the causative bacteria and their susceptibility. However, defining appropriate antimicrobial therapy directed to the causative bacteria in DFO is challenging since it requires bone biopsy (BB) procedures which are underused in clinical practice for various reasons: lack of availability, cost, and delay. Some clinicians also find bone biopsy cumbersome or too invasive.

To overcome these barriers, we have set up for a few years a bedside blind BB procedure performed by diabetologists at the bedside in the clinical ward. Since then, this method has been used in more than 200 patients with DFO in the diabetology departments of Lariboisiere Hospital and Bichat Hospital (Paris). We have recently published our observational data of 79 patients showing that bedside BB is a simple, safe and efficient procedure for the diagnosis of DFO with a similar rate of complete healing at 12 months compared to conventional surgical or radiological bone biopsies. In order to extend and confirm these preliminary and observational results, the aim of this study is to compare the efficiency and safety of bedside BB versus conventional bone biopsy in a randomized controlled trial (RCT) of patients with DFO. Our hypothesis is that bedside BB is non-inferior to conventional bone biopsy in DFO and can be used as a simpler alternative procedure to document DFO

DETAILED DESCRIPTION:
During their lifetime, 15 to 25% of patients with diabetes mellitus will develop a Diabetic Foot Ulcer (DFU) related to neuropathy and/or peripheral arterial disease1. DFU is the leading cause of non-traumatic lower-extremity amputation worldwide. DFO, which complicates up to 60% of DFU, is a major trigger of amputation in over 80% of persons with diabetes resulting in subsequent loss of quality of life2. It has been shown that medical treatment of DFO may prevent amputations with early diagnosis of osteomyelitis and appropriate use of antibiotics3. Empirical antimicrobial treatment is not recommended for DFO as for other chronic infections. Surgically or radiologically acquired bone sample for culture is the reference standard recommended by the International Working Group of Diabetic Foot (IWGDF) to diagnose DFO and to determine the causative bacteria and their susceptibility4. However, defining appropriate antimicrobial therapy directed to the causative bacteria in DFO is challenging since it requires bone biopsy (BB) procedures which are underused in clinical practice for various reasons including lack of availability, cost, and delay. Some clinicians also find bone biopsy cumbersome or too invasive.

To overcome these barriers, we have set up for a few years a bedside blind BB procedure performed by a physician at the bedside in the clinical ward. Since then, this method has been used in more than 200 patients with DFO in the diabetology departments of Lariboisiere Hospital and Bichat Hospital (Paris). We have recently published our observational data of 79 patients showing that bedside BB is a simple, safe and efficient procedure for the diagnosis of DFO with a similar rate of complete DFU healing at 12 months compared to conventional surgical or radiological bone biopsies6. In order to extend and confirm these preliminary and observational results, the aim of this study is to compare the efficiency and safety of bedside versus conventional BB in a randomized controlled trial (RCT) of patients with DFO. Our hypothesis is that bedside BB is non inferior to conventional BB in DFO outcomes and can be used as a simpler alternative procedure to document DFO.

The main objective is to demonstrate non-inferiority of beside blind bone biopsy compared to conventional bone biopsy (surgical or radiological) on DFO remission without surgery at 1 year.

The secondary objectives of this study are to:

1. compare clinical efficacy between groups of bone biopsy
2. compare microbiological culture results between groups
3. compare the safety of both procedures
4. compare DFO remission according to results of BB (negative or positive)

The health economic of this study are to:

1. to estimate total costs for the intervention and total medical costs in each groups
2. to estimate total quality adjusted life years (QALYs) based upon EQ5D5L scores
3. to calculate the point estimate of the incremental cost utility ratio and estimate the probability of decremental cost effectiveness for the beside blind bone biopsy compared to conventional biopsy.

In this study, we will include subjects with diabetes and DFU with a suspicion of DFO. DFO is a complication of a large amount of DFU and is a major trigger of lower limb amputations. As we will include participants before bacteriological confirmation of DFO through bone biopsy, we will use the clinical and radiological criteria for DFO according to IWGDF 2019 guidelines4.

These criteria include having at least one of the following signs:

* A positive probe to bone test and abnormalities on plain X-ray suggestive for osteomyelitis
* Signs of osteomyelitis on CT-scan and/or MRI and/or white blood cell SPECT/CT and/or 18Fluor-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose-positron emission tomography (FDG-PET)/CT- scan

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study must fulfill all of the following criteria:

* Aged >18 years
* Diabetes mellitus
* At least one of the following signs of osteomyelitis according to IWGDF 2019 guidelines:

A positive probe to bone test and abnormalities on plain X-ray suggestive for osteomyelitis Signs of osteomyelitis on CT-scan and/or MRI and/or white blood cell SPECT/CT and/or FDG-PET/CT-scan

- Absence of antibacterial therapy within 14 days before inclusion

Exclusion Criteria:

Patients fulfilling any of the following criteria are not eligible for inclusion in this study:

* Urgent need for surgery
* Critical limb ischemia which cannot be corrected by revascularization procedure
* Subjects that (are likely to) undergo surgical or percutaneous revascularization are not excluded
* Antibiotic treatment in the last 15 days before bone biopsy
* Osteomyelitis in the area of the Charcot foot destructive process
* Unlikely to live at least 1 year
* Not being able to give informed consent and willing to comply with the research protocol
* Pregnant or breastfeeding women
* Absence of affiliation to French social insurance
* State medical aid (AME)
* Deprivation of liberty, being under a legal protective measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
the remission of DFO | 12 months
  The remission of DFO at 12 months and is defined by a composite criterion as:
  * an epithelialized ulcer for 28 consecutive days
  * and absence of local inflammation and/or stabilization or improvement of radiologic abnormalities
  * and no need for surgery of the foot to treat DFO during follow-up

SECONDARY OUTCOMES:
Clinical efficacy | 12 months
  Remission of DFO at 6 months
Clinical efficacy | 12 months
  Need for surgery for initial DFU during follow-up
Clinical efficacy | 12 months
  Recurrence of DFU during follow-up
Clinical efficacy | 12 months
  Death during follow-up
Clinical efficacy | 12 months
  Number of hospitalizations
Clinical efficacy | 12 months
  length of hospitalizations
Clinical efficacy | 12 months
  Length of stay of the initial hospitalization (in days)
Microbiological results | 12 months
  Number of microorganisms per biopsy
Microbiological results | 12 months
  Number of resistant microorganisms per biopsy
Microbiological results | 12 months
  Total duration of the antibacterial therapy (mean in days)
Occurrence of adverse events during the study | 12 months
Remission rate of DFO | 12 months
  Remission rate of DFO at 12 months according to microbiological results of BB (positive or negative)
costs: Average costs of the biopsies | 1 month
costs: Average total 1-year costs | 12 months
Average 1 year QALY | 12 months
Incremental cost effectiveness ratio | 12 months
  defined as the difference in average total costs/ average total QALY

CONTACTS AND LOCATIONS:
Overall Officials: Louis Potier, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Bichat - Claude Bernard Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided